CLINICAL TRIAL: NCT00734500
Title: Anidulafungin PK in Infants and Toddlers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Cohen-Wolkowiez (Other)
Responsible Party: Sponsor-Investigator, Michael Cohen-Wolkowiez, Assistant Professor, Department of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000637
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Results first posted 2011-12-14 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Invasive Fungal Infections
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Anidulafungin

ARMS (1):
- Treatment (Experimental): Treatment
  Interventions: Drug: Anidulafungin

INTERVENTIONS:
Drug: Anidulafungin — Intravenous form. Loading Dose: 3 mg/kg/dose. Maintenance dose: 1.5 mg/kg/dose. Treatment duration: 5 days total.
  Other Names: Eraxis

SUMMARY:
This is a prospective, open-label, single center, pharmacokinetic study of anidulafungin in infants and toddlers less than 24 months of age with suspected serious infection. There will be up to 24 subjects enrolled; each will receive anidulafungin. Patients will receive anidulafungin 3 mg/kg loading dose on day 1 of study and will receive 1.5 mg/kg every 24 hours on study days 2-5.Plasma pharmacokinetics will be evaluated using a limited sampling scheme. We hypothesize that the PK parameters of anidulafungin will not differ from those observed in older children and adults.

ELIGIBILITY:
Inclusion Criteria:

* Age < 24 months at the time of enrollment
* Patient must have sufficient venous access to permit administration of study medication
* Infant or toddler suspected to have a serious infection and from whom a blood culture has been obtained with 48 hours of study entry
* Availability and willingness of the parent/legally authorized representative to provide written informed consent.

Exclusion Criteria:

* Patients with a history of anaphylaxis attributed to an echinocandin
* Any other concomitant condition, which in the opinion of the investigator would preclude a patient's participation in the study
* Previous participation in this study
* Previous exposure to an echinocandin in the month prior to study.

Ages: 48 Hours to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Anidulafungin: Intravenous anidulafungin (loading dose, 3 mg/kg once followed by 1.5 mg/kg/day)
Period: Overall Study
Arm/Group | Anidulafungin
Started | 15
Completed | 14
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Anidulafungin
Number analyzed (Participants) | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 0.22 (0.32)
Age, Customized [Number; unit: participants]
  <=24 months | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: The Pharmacokinetics (Area Under the Curve) of Anidulafungin in Infants and Toddlers Less Than 24 Months of Age With Suspected Serious Infection.
Description: Area under the curve at steady state
Time Frame: 5 days
Measure: Median (Full Range); unit: µg*h/mL
Arm/Group | Anidulafungin
Number analyzed (Participants) | 14
µg*h/mL | 84 [30 to 278]

2. Secondary Outcome: Safety (Participants With Adverse Events) of Anidulafungin in Infants and Toddlers Less Than 24 Months of Age With Suspected Serious Infection.
Description: Participants with Adverse events were collected during the study drug administration phase up to 10 days after last dose of study drug.
Time Frame: During and up to 10 days after last dose of study drug.
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 15
participants | 8

ADVERSE EVENTS:
Arm/Group | Anidulafungin
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 2/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anidulafungin (N=15)
Death (Cardiac disorders) | 1 (1) — Cardiac and respiratory failure - family withdrew care - patient died soon after administration of 1st dose of study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anidulafungin (N=15)
Direct hyperbilirubinemia (Gastrointestinal disorders) | 2 (2) — 2 subjects experienced direct hyperbilirubinemia possibly related to study drug; study drug was stopped in 1 of these patients. Both patients had history of previous hyperbilirubinemia episodes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No